CLINICAL TRIAL: NCT06209944
Title: A Retrospective Review on Charlson Comorbidity Index (CCI) as a Predictor of Return-of-spontaneous-circulation and Survival-to-discharge of Geriatric In-hospital Cardiopulmonary Resuscitation (CPR) in a Regional Acute Hospital in Hong Kong
Brief Title: Charlson Comorbidity Index and Outcome of Cardiopulmonary Resuscitation in Geriatric Patients in Hong Kong
Status: Completed | Type: Observational
Sponsor: Jane Yidan Zhu (Other)
Responsible Party: Sponsor-Investigator, Jane Yidan Zhu, Dr Jane Yidan Zhu, Associate Consultant, Haven of Hope Hospital
Organization: Haven of Hope Hospital (Other)
Other Study IDs: CCI and outcome of CPR
Record Dates: First submitted 2023-10-01; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Comorbidities and Coexisting Conditions; Cardiopulmonary Resuscitation; Geriatrics
MeSH Terms: interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiopulmonary resuscitation — cardiac compression, endotracheal intubation, defibrillation, and use of cardiovascular medications, to restore circulation in patients with cardiac arrest

SUMMARY:
The goal of this observational study is to learn about the factors affecting the outcome (survival) of cardiopulmonary resuscitation in older persons in a hospital. The main questions it aims to answer are:

* Whether age would affect outcome
* Whether Charlson Comorbidity Index would affect outcome
* Whether the conditions (e.g. heart rhythm) immediately before resuscitation would affect survival.

Researchers would compare the patients who deceased with the patients who survived.

DETAILED DESCRIPTION:
The goal of this review was to investigate the impact of age, existing medical conditions. and other factors before cardiac arrest in predicting outcome of in-hospital cardiopulmonary resuscitation (CPR) of older persons.

It was conducted on all patients aged ≥ 65, who underwent CPR in acute medical and geriatric wards (excluding Intensive Care Unit) in United Christian Hospital from January 2017 to December 2018.

ELIGIBILITY:
Inclusion Criteria:

* All adults aged 65 or above with in-hospital cardiac arrest and undergoing CPR in wards of Department of Medicine and Geriatrics (excluding Intensive Care Unit (ICU)) in United Christian Hospital (total bed 1,174 with 16 ICU beds) in Hong Kong from 1 January 2017 to 31 December 2018
* In patients with multiple resuscitation events, only the first in-hospital CPR was included.

Exclusion Criteria:

* Patients with existing Do-Not-Attempt-Cardiopulmonary-Resuscitation (DNACPR) order
* Patients younger than 65 years old
* Out-of-hospital CPR in the index admission
* CPR occurred in ICU / Emergency Department / Operating Theatre / wards other than medical wards

Ages: 65 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All adults aged 65 or above with in-hospital cardiac arrest and undergoing CPR in wards of Department of Medicine and Geriatrics (excluding Intensive Care Unit (ICU)) in United Christian Hospital (a regional acute hospital with total bed 1,174 with 16 ICU beds) in Hong Kong from 1 January 2017 to 31 December 2018
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
sustained return of spontaneous circulation (ROSC), survival at 24 hours, survival at hospital discharge, and at 1 year. | 2017 - 2018
  Sustained ROSC is defined as documented return of adequate circulation in the absence of ongoing chest compressions, and the duration should be of 20 minutes or above

CONTACTS AND LOCATIONS:
Overall Officials: JANE YIDAN ZHU, Principal Investigator — Haven of Hope Hospital, Hong Kong
Locations (1):
- Haven of Hope Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT06209944/Prot_SAP_000.pdf